CLINICAL TRIAL: NCT06360393
Title: Inhaler Adherence and Inhalation Technique Assessed by a Smart Spacer in Patients with Severe Asthma on Biologics
Acronym: OUTERSPACE-3
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Trudell Medical International (Industry)
Responsible Party: Sponsor
Other Study IDs: 17384
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: Severe asthma; Biologics; Digital home monitoring; Digital spacer; Adherence; Inhalation technique
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe asthma patients on biologics: Participants diagnosed with severe asthma using a biologic medication and medium or high dose ICS + LABA with or without LAMA and/or SABA via pMDI and spacer. Participants are being treated at one of the five severe asthma clinics in The Netherlands.
  Interventions: Device: Smart spacer

INTERVENTIONS:
Device: Smart spacer — Participants' inhalation medication adherence and inhalation technique will be monitored using a smart spacer. Their usual medication regime will be continued and they will not receive information about their adherence or inhalation technique measured by the spacer during the follow-up year (except for any interventions that will be done in standard care).

SUMMARY:
Severe refractory asthma affects about 3.5% of asthma patients, often necessitating biologic therapy in addition to standard treatment. However, little is understood about maintenance and reliever inhalation medication adherence in these cases which might impact overall biologic response. Objectively monitoring inhalation medication adherence remains a significant challenge. The Smart AeroChamber® device, capable of measuring adherence and inhalation technique, is untested in severe asthma patients on biologics, presenting a potentially cost-effective solution to monitor adherence and better understand treatment response.

This study aims to assess the feasibility of the Smart AeroChamber® device in severe asthma patients on biologic therapy, with objectives to:

1. Evaluate inhalation medication adherence patterns and inhaler technique, and comparing that adherence data with traditional measures e.g. the Test of Adherence to Inhalers (TAI), and an inhalation technique checklist.
2. Investigate the association between inhaled medication adherence and clinical outcomes such as exacerbations, short-acting beta-agonists (SABA) use, oral corticosteroids use (OCS), Fractional Exhaled Nitric Oxide (FeNO), blood eosinophil count, and Asthma Control Questionnaire (ACQ) scores.
3. Assess patient and healthcare provider satisfaction and usability of the Smart AeroChamber® device.

The study design is prospective and observational, with a sample size of 110 adult patients diagnosed with severe asthma using biologic therapy. Participants will be followed for 12 months, during which they will receive Smart AeroChamber® devices. These devices will measure medication adherence and inhaler technique, and undergo assessments of clinical outcomes at regular intervals. Usability and satisfaction will also be evaluated using the Systems Usability Scale (SUS) in patients and healthcare professionals.

The study will be conducted across five severe asthma clinics in the Netherlands. Data analysis will involve comparing the inhalation medication adherence data with traditional measures for adherence and inhalation technique, assessing clinical outcomes, and evaluating usability and satisfaction. The findings from this study will provide insights into the feasibility and effectiveness of using digital devices like the Smart AeroChamber® to support medication adherence and possibly improve outcomes in patients with severe asthma on biologic therapy.

DETAILED DESCRIPTION:
Rationale:

Despite the availability of effective inhaled medications, 15% of asthma patients remain uncontrolled on medium to high dose inhaled corticosteroids (ICS) and LABA, comprising difficult-to-treat asthma and severe refractory asthma groups. GINA guidelines stress the importance of assessing adherence and technique before step-up treatment due to associated risks and costs.

Research underscores the efficacy and cost-effectiveness of investing in adherence and technique support, particularly in this population. However, there is limited understanding of ICS adherence during biologic therapy, despite its increasing use. Studies on biologics like mepolizumab suggest associations between ICS adherence and improved outcomes, while data on others like benralizumab are less conclusive.

Indeed, non-adherence and poor technique is widely reported in patients with all severities of asthma and is associated with increased morbidity and economic burden. Objectively assessing and enhancing adherence remains one of the major challenges for physicians, pharmacists and nurses. Limited studies on digital tools for adherence management exist, particularly for pMDIs in combination with spacers. Digital technologies are promising in addressing these challenges, but studies on devices capable of objectively measuring adherence and technique, especially in patients using pMDIs, are lacking. The Smart AeroChamber® device presents an innovative solution, showing potential in clinical trials for asthma and COPD. The Smart AeroChamber® is a CE-certified device. However, its application in severe asthma patients on biologics remains unexplored, presenting an opportunity to enhance adherence support and treatment outcomes in this cost-sensitive population.

The aim:

This study aims to evaluate the feasibility of using a Smart Spacer device in patients with severe asthma who are on biologic therapy. The research aims to achieve several objectives:

1. Assess medication adherence patterns and inhaler technique using the Smart Spacer device and compare the data with traditional adherence measures, such as the Test of Adherence to Inhalers (TAI), and an inhalation technique checklist.
2. Evaluate the association between adherence measured by the Smart Spacer device and various clinical outcomes including exacerbations, use of short-acting beta agonists (SABA) and oral corticosteroids (OCS), Fractional exhaled Nitric Oxide (FeNO) results, blood eosinophil count, and asthma control questionnaire (ACQ) scores.
3. Assess the usability and satisfaction of patients and healthcare providers with the Smart Spacer device, using the System Usability Scale (SUS).

Study Design:

This study adopts a prospective, observational design.

Inclusion Criteria:

Participants eligible for inclusion are adults aged over 18 years, diagnosed with severe asthma by a physician according to GINA guidelines. They must be using a biologic medication (omalizumab, mepolizumab, reslizumab, benralizumab, dupilumab or tezepelumab) and medium or high dose ICS + LABA with or without LAMA and/or SABA via pMDI in combination with a spacer. Additionally, participants must be willing to provide informed consent.

Exclusion Criteria:

Participants are excluded from participation when they are unable to sufficiently understand and read the Dutch language, being pregnant or being terminally ill.

Sample Size:

The study aims to include a total of 110 patients.

Setting:

The study is conducted in five severe asthma clinics across various regions of the Netherlands (Medical Center Leeuwarden, Martini Hospital Groningen, Isala Zwolle, Sint Franciscus Gasthuis, and University Medical Centrer Groningen).

Baseline Assessment:

Participants undergo characterization during an intake visit to the severe asthma clinic, including demographic data, medical history, spirometry tests, FeNO measurement, blood eosinophil count, ACQ assessment, adherence evaluation using TAI, and inhaler technique assessment via checklist. Subsequently, participants receive two fully charged smart spacers, one for each period of three months, along with instructions for use.

Follow-up:

After 4 weeks, participants are contacted to check the functionality of the smart spacer and receive assistance if needed. A follow-up call at 3-months and 9-months into the study remind participants to switch to the next smart spacer. A physical visit is scheduled at the 6-month mark for further assessment, including ACQ administration and collection of smart spacers for replacement.

End of Study Assessment:

At the end of the 12-month study period, participants undergo a final physical visit for assessment of various parameters including FeNO, blood eosinophil count, lung function, ACQ score, inhaler technique, and documentation of exacerbations and OCS use. Smart spacer data analysis is conducted centrally, and feedback is provided to study sites. Additionally, usability and satisfaction surveys are completed by patients and study nurses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Confirmed asthma diagnoses (≥12% and >200 ml reversibility in FEV1 or positive histamine/methacholine provocation test or FeNO ≥50) according to the asthma guidelines
* Diagnosed with severe, refractory asthma with eligibility for treatment with specific asthma biologics (omalizumab, mepolizumab, benralizumab, reslizumab, dupilumab)
* Using medium or high ICS + LABA +/- LAMA+/-SABA) by pMDI+spacer
* Willing to sign informed consent

Exclusion Criteria:

* The use of the Symbicort Aerosol or the Trixeo Aerosphere in combination with a spacer (these inhalers are not compatible with the smart spacer)
* Inability to sufficiently understand and read the Dutch language
* Current pregnancy
* Currently terminally ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged over 18 years, diagnosed with severe asthma by a physician according to GINA guidelines. They must be using a biologic medication (omalizumab, mepolizumab, reslizumab, benralizumab, or dupilumab) and medium or high dose ICS + LABA with or without LAMA and/or SABA via pMDI and spacer.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparative analysis of smart spacer medication adherence and inhaler technique against Test of Adherence to Inhalers (TAI-12) | TAI is measured at baseline and 12 months
  An evaluation of the inhalation adherence patterns and inhaler techniques of patients utilizing smart spacer devices in comparison to traditional inhaler usage assessed by the Test of Adherence to Inhalers (TAI-12).
  TAI is a questionnaire which identifies patients with low adherence, determines the degree of adherence and gives an idea of the type or pattern of non-compliance. The TAI-12 consists of 10 questions for the patient and 2 questions for the healthcare provider and identifies patients with poor adherence and their degree of adherence. The scoring for the patient part is: for each question ranges from 1 to 5 (1 = worst compliance to 5 = best compliance). All items provide a total score of between 10 (minimum) and 50 (maximum). A higher score is related to better adherence. The scoring of the healthcare provider part is: a minimum of 2 points and a maximum of 4 points. A higher score also relates to a better adherence.
Comparison of smart spacer medication adherence patterns (adherence and inhaler technique) with inhaler checklist examined by pulmonologist or pulmonary nurse | Inhaler checklist is assessed at baseline and 12 months
  An evaluation of the inhalation adherence patterns and inhaler techniques of patients utilizing smart spacer devices in comparison to traditional inhaler usage assessment by healthcare professionals using an inhalation technique checklist.
  The inhalation technique checklist is created by following the national inhalation technique guidelines by the Lung Foundation in The Netherlands (Long Alliantie Nederland, LAN), specifically for using a pMDI in combination with a spacer. The checklist consists of 8 points to assess the inhalation technique on (from the preparation of the device, to the positioning of the device and posture of the patient, and the actual inhalation).

SECONDARY OUTCOMES:
Assessing the association of smart spacer assessed adherence with annual exacerbation rate | Over a period of 12 months
  An assessment of the association between inhalation medication adherence measured by smart spacer devices and the annual exacerbation rate.
  The annual exacerbation rate will include the number of exacerbations of the participant in the one-year follow-up and the severity of the exacerbation (e.g. increased reliever use, oral corticosteroid use, emergency room visit, hospitalization).
Assessing the association of smart spacer assessed adherence with reliever inhaler use (e.g. SABA) | Over a period of 12 months
  An examination of the possible association between inhalation medication adherence measured by smart spacer devices and the use of reliever medication.
  The use of reliever medication will also be monitored by the smart spacer and it is included as a question in the Asthma Control Questionnaire (question 6).
Assess the association of smart spacer assessed adherence with oral corticosteroids use | Over a period of 12 months
  An examination of the possible association between inhalation medication adherence measured through smart spacer devices and the use of oral corticosteroids (OCS).
  The use of OCS will be defined as total annual OCS exposure (in milligrams) as well as the number of high dose (> 30 milligrams) short courses (between 3 to 14 days).
Assess the association of smart spacer assessed adherence with FeNO results | FeNO is measured at baseline and 12 months
  An examination of the possible association between inhalation medication adherence measured through smart spacer devices and FeNO measurements.
  Fractional exhaled nitric oxide (FeNO) serves as an indicator of inflammation in asthma. It has been employed as a measure to detect non-compliance with inhaled corticosteroid (ICS) therapy. Individuals who do not adhere to ICS treatment typically exhibit elevated FeNO levels since ICS effectively suppress FeNO. A high FeNO level despite ICS usage suggests ongoing inflammation in the airways due to asthma, increasing the likelihood of exacerbations. The difference in FeNO measured at baseline and 12 months will be compared the overall ICS adherence.
Assess the association of smart spacer assessed adherence with blood eosinophils | Blood eosinophils measured at baseline and 12 months
  An examination of the possible association between inhalation medication adherence measured through smart spacer devices and blood eosinophils.
  Blood eosinophils are a type of white blood cell that plays a significant role in the immune response, particularly in allergic reactions and inflammatory conditions. Asthma is characterized by chronic inflammation of the airways, and eosinophils are one of the key inflammatory cells involved. Elevated levels of eosinophils in the blood can indicate ongoing inflammation in the airways. Blood eosinophil levels can also serve as a biomarker for predicting response to certain asthma treatments, particularly corticosteroids. Elevated blood eosinophil levels have been associated with an increased risk of asthma exacerbations. The difference in eosinophils measured at baseline and 12 months will be compared the overall ICS adherence.
Assess the association of smart spacer assessed adherence with asthma control (ACQ-6) | ACQ is measured at baseline, 6 months and 12 months
  An examination of the possible association between adherence measured through smart spacer Asthma Control assessed with the Asthma Control Questionnaire (ACQ-6).
  This questionnaire consists of six questions about the severity of symptoms which a patient experiences. The score range per question is 0 to 7 (0 = never and 7 = always). The total score will be calculated by dividing the sum of all scores by the amount of questions. A higher score is associated with worse asthma control. The difference in ACQ outcomes at baseline, 6-months and 12 months will be compared the overall ICS adherence.
Assess the association of smart spacer assessed adherence with spirometry results | Spirometry is performed at baseline and 12 months
  An examination of the possible association between adherence measured through smart spacer devices and spirometry results.
  Spirometry is a pulmonary function test that measures how much air a person can inhale and exhale, as well as how quickly they can exhale. Asthma often shows a reduced forced expiratory volume in one second (FEV1) and a reduced FEV1 to forced vital capacity (FVC) ratio, indicating obstruction. Lower spirometry readings, particularly a lower FEV1, may indicate poorly controlled asthma, which is associated with an increased risk of exacerbations. Measured: Forced Vital Capacity (FVC) (% pred), Forced Expiratory Volume in one second (FEV1) (% pred), Peak Expiratory Flow (PEF) (L/min), and FEV1/FVC ratio. The difference in spirometry results at baseline and 12 months will be compared the overall ICS adherence.

OTHER OUTCOMES:
Assess usability and patient satisfaction using the System Usability Scale | SUS is measured at 12 months
  The usability and patient satisfaction will be measured using the System Usability Scale (SUS).
  The SUS provides a simple and standardized effective tool for assessing usability and patient satisfaction with healthcare technologies. The SUS consists of ten statements related to usability, with respondents asked to rate their level of agreement with each statement on a five-point Likert scale ranging from "Strongly Disagree" (1 point) to "Strongly Agree" (5 points).
  The score for the five odd-numbered questions is determined by subtracting 1 from the scored points (X-1). The score for the five even-numbered questions is calculated by deducting the scored points from 5 (5-X). By adding up these two scores and multiplying the total by 2.5, the SUS score is calculated. The total scores range from 0 to 100. Higher scores indicate better usability, with scores above 70 considered above average and scores above 80 indicating excellent usability.
Assess usability and healthcare provider satisfaction using the System Usability Scale | SUS is measured at 12 months
  The usability and healthcare provider satisfaction will be measured using the System Usability Scale (SUS).
  The SUS provides a simple and standardized effective tool for assessing usability and healthcare providers' satisfaction with healthcare technologies. The SUS consists of ten statements related to usability, with respondents asked to rate their level of agreement with each statement on a five-point Likert scale ranging from "Strongly Disagree" (1 point) to "Strongly Agree" (5 points).
  The score for the five odd-numbered questions is determined by subtracting 1 from the scored points (X-1). The score for the five even-numbered questions is calculated by deducting the scored points from 5 (5-X). By adding up these two scores and multiplying the total by 2.5, the SUS score is calculated. The total scores range from 0 to 100. Higher scores indicate better usability, with scores above 70 considered above average and scores above 80 indicating excellent usability.

CONTACTS AND LOCATIONS:
Overall Officials: Job FM van Boven, PharmD, PhD, Principal Investigator — University Medical Center Groningen
Locations (5):
- Netherlands (5):
  - Isala, Zwolle, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Foundation Martini Hospital, Groningen, Provincie Groningen
  - Stichting Sint Franciscus Vlietland Groep, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hekking PW, Wener RR, Amelink M, Zwinderman AH, Bouvy ML, Bel EH. The prevalence of severe refractory asthma. J Allergy Clin Immunol. 2015 Apr;135(4):896-902. doi: 10.1016/j.jaci.2014.08.042. Epub 2014 Oct 16. PMID 25441637
- [Background] McQueen RB, Sheehan DN, Whittington MD, van Boven JFM, Campbell JD. Cost-Effectiveness of Biological Asthma Treatments: A Systematic Review and Recommendations for Future Economic Evaluations. Pharmacoeconomics. 2018 Aug;36(8):957-971. doi: 10.1007/s40273-018-0658-x. PMID 29736895
- [Background] Barry LE, Sweeney J, O'Neill C, Price D, Heaney LG. The cost of systemic corticosteroid-induced morbidity in severe asthma: a health economic analysis. Respir Res. 2017 Jun 26;18(1):129. doi: 10.1186/s12931-017-0614-x. PMID 28651591
- [Background] Hale EM, Greene G, Mulvey C, Mokoka MC, van Boven JFM, Cushen B, Sulaiman I, Brennan V, Lombard L, Walsh J, Plunkett S, McCartan TA, Kerr PJ, Reilly RB, Hughes C, Kent BD, Jackson DJ, Butler M, Counihan I, Hayes J, Faul J, Kelly M, Convery R, Nanzer AM, Fitzgerald JM, Murphy DM, Heaney LG, Costello RW; INCA Research Team. Use of digital measurement of medication adherence and lung function to guide the management of uncontrolled asthma (INCA Sun): a multicentre, single-blinded, randomised clinical trial. Lancet Respir Med. 2023 Jul;11(7):591-601. doi: 10.1016/S2213-2600(22)00534-3. Epub 2023 Mar 21. PMID 36963417
- [Background] d'Ancona G, Kavanagh J, Roxas C, Green L, Fernandes M, Thomson L, Dhariwal J, Nanzer AM, Jackson DJ, Kent BD. Adherence to corticosteroids and clinical outcomes in mepolizumab therapy for severe asthma. Eur Respir J. 2020 May 7;55(5):1902259. doi: 10.1183/13993003.02259-2019. Print 2020 May. PMID 32060061
- [Background] d'Ancona G, Kavanagh JE, Dhariwal J, Hearn AP, Roxas C, Fernandes M, Green L, Thomson L, Nanzer AM, Jackson DJ, Kent BD. Adherence to inhaled corticosteroids and clinical outcomes following a year of benralizumab therapy for severe eosinophilic asthma. Allergy. 2021 Jul;76(7):2238-2241. doi: 10.1111/all.14737. Epub 2021 Jan 26. No abstract available. PMID 33432682
- [Background] Dekhuijzen R, Lavorini F, Usmani OS, van Boven JFM. Addressing the Impact and Unmet Needs of Nonadherence in Asthma and Chronic Obstructive Pulmonary Disease: Where Do We Go From Here? J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):785-793. doi: 10.1016/j.jaip.2017.11.027. Epub 2018 Jan 12. PMID 29339126
- [Background] van Boven JF, Ryan D, Eakin MN, Canonica GW, Barot A, Foster JM; Respiratory Effectiveness Group. Enhancing Respiratory Medication Adherence: The Role of Health Care Professionals and Cost-Effectiveness Considerations. J Allergy Clin Immunol Pract. 2016 Sep-Oct;4(5):835-46. doi: 10.1016/j.jaip.2016.03.007. PMID 27587317
- [Background] O'Dwyer S, Greene G, MacHale E, Cushen B, Sulaiman I, Boland F, Bosnic-Anticevich S, Mokoka MC, Reilly RB, Taylor T, Ryder SA, Costello RW. Personalized Biofeedback on Inhaler Adherence and Technique by Community Pharmacists: A Cluster Randomized Clinical Trial. J Allergy Clin Immunol Pract. 2020 Feb;8(2):635-644. doi: 10.1016/j.jaip.2019.09.008. Epub 2019 Sep 27. PMID 31568927
- [Background] Jansen EM, van de Hei SJ, Dierick BJH, Kerstjens HAM, Kocks JWH, van Boven JFM. Global burden of medication non-adherence in chronic obstructive pulmonary disease (COPD) and asthma: a narrative review of the clinical and economic case for smart inhalers. J Thorac Dis. 2021 Jun;13(6):3846-3864. doi: 10.21037/jtd-20-2360. PMID 34277075
- [Background] Vincken W, Levy ML, Scullion J, Usmani OS, Dekhuijzen PNR, Corrigan CJ. Spacer devices for inhaled therapy: why use them, and how? ERJ Open Res. 2018 Jun 18;4(2):00065-2018. doi: 10.1183/23120541.00065-2018. eCollection 2018 Apr. PMID 29928649
- [Background] Price DB, Roman-Rodriguez M, McQueen RB, Bosnic-Anticevich S, Carter V, Gruffydd-Jones K, Haughney J, Henrichsen S, Hutton C, Infantino A, Lavorini F, Law LM, Lisspers K, Papi A, Ryan D, Stallberg B, van der Molen T, Chrystyn H. Inhaler Errors in the CRITIKAL Study: Type, Frequency, and Association with Asthma Outcomes. J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):1071-1081.e9. doi: 10.1016/j.jaip.2017.01.004. Epub 2017 Mar 9. PMID 28286157
- [Background] Normansell R, Kew KM, Mathioudakis AG. Interventions to improve inhaler technique for people with asthma. Cochrane Database Syst Rev. 2017 Mar 13;3(3):CD012286. doi: 10.1002/14651858.CD012286.pub2. PMID 28288272
- [Background] Dierick BHJ, Achterbosch M, Been-Buck S, Klemmeier T, van de Hei SJ, Hagedoorn P, Kerstjens HAM, Kocks JWH, van Boven JFM. Can electronic monitoring with a digital smart spacer support personalised medication adherence and inhaler technique education in patients with asthma?: Protocol of the randomised controlled OUTERSPACE trial. BMJ Open. 2022 Jun 13;12(6):e059929. doi: 10.1136/bmjopen-2021-059929. PMID 35697450
- [Background] Dierick BJH, Been-Buck S, Klemmeier T, Hagedoorn P, van de Hei SJ, Kerstjens HAM, Kocks JWH, Zijp TR, Wessels AMA, Touw DJ, van Boven JFM. Digital spacer data driven COPD inhaler adherence education: The OUTERSPACE proof-of-concept study. Respir Med. 2022 Sep;201:106940. doi: 10.1016/j.rmed.2022.106940. Epub 2022 Jul 31. PMID 35933835
- [Background] Eikholt AA, Wiertz MBR, Hew M, Chan AHY, van Boven JFM. Electronic monitoring devices to support inhalation technique in patients with asthma: A Narrative Review. Curr Treat Options Allergy. 2023; 10:28-52 doi: 10.1007/s40521-023-00328-7.